CLINICAL TRIAL: NCT05000528
Title: Etude Pilote d'évaluation de l'efficacité de l'ETP Sur l'Insomnie Chronique
Brief Title: Evaluation of the Effectiveness of Patient Therapeutic Education on Chronic Insomnia
Acronym: ETP-INSOMNIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2020-2/BA-1
Record Dates: First submitted 2021-07-22; First posted 2021-08-11 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic education (Experimental)
  Interventions: Other: therapeutic education; Other: Actimetry
- Individualized consultation (Active Comparator)
  Interventions: Other: Actimetry

INTERVENTIONS:
Other: therapeutic education — In groups of 5-6, patients will have a one-day therapeutic training session comprising 4 workshops: how to create a sleep agenda; normal sleep; sleep hygiene; medical treatments.
  Arms: Therapeutic education
Other: Actimetry — once from inclusion for 2 weeks, second for 2 weeks starting 2 weeks after intervention

SUMMARY:
20 to 30% of the general population suffers from chronic insomnia. Cognitive behavioral therapy (CBT) is the first-line treatment, but unfortunately its implementation is complex. Long waiting times for a consultation / exploration, too short a consultation period, non-reimbursement of specialists and a lack of trained staff make the current care of insomniac patients difficult. Patients are thus treated late, often with heavy drug treatment, dependence on sleeping pills, difficult withdrawal and / or reactive mood disorders. The treatment is therefore limited to advice on sleep hygiene and a restriction of time spent in bed without ultimately intervening in the cognitive domain. Therapeutic education consists of empowering the patient in the management of chronic insomnia through group education workshops. The patient learns the principles of normal sleep, the way in which sleep evolves with aging, the dangers of treatments as well as the rules of sleep hygiene and the behaviors to modify to sleep well. In addition to benefiting from sharing of experience with other patients, therapeutic education makes the care pathway smoother and considerably reduces the long waiting times of the traditional care pathway in consultation.

The study investigators hypothesize that therapeutic education is more effective as a treatment for chronic insomnia than traditional management in individualized consultation (IC). Thus, therapeutic education could constitute an effective alternative to CBT.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent
* The patient must be a member or beneficiary of a health insurance plan
* Patient must understand and read French
* Patient with ICSD-3 diagnostic criteria for chronic insomnia: ISI score > 14/28.

Exclusion Criteria:

* Patient with cognitive impairment as assessed by the investigator
* Patient with shift work
* Patients scoring > 10/24 on the Epworth sleepiness scale
* Patient suffering from medical or psychiatric illnesses which may, in the opinion of the investigator, compromise the subject's state of health or ability to participate in the study.
* Patient with chronic alcohol consumption or drug abuse
* Patient unable to express consent.
* Pregnant, parturient or breastfeeding patient.
* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Improvement in chronic insomnia between groups | Day 28
  Change in Insomnia Severity Index (ISI) score (Score between 0 - 28) from inclusion

SECONDARY OUTCOMES:
Change in total sleeping time between groups | Day 28
  Change in total sleeping time (minutes) from inclusion
Change in time in bed between groups | Day 28
  Change in time in bed (minutes) from inclusion
Change in effective sleep | Day 28
  Time between going to bed and falling asleep (minutes). Average time for the 2 weeks following inclusion versus the 2 weeks preceding the study end measured by actimetry bracelet
Change in sleep latency | Day 28
  % total sleeping time / time in bed. Average time for the 2 weeks following inclusion versus the 2 weeks preceding the study end measured by actimetry bracelet
Change in intra-sleep time | Day 28
  Change in time between going to bed and falling asleep (minutes) since inclusion, data collected from patient sleep agenda
Change in anxiety since baseline between groups | Day 28
  State-Trait Anxiety Inventory (STAI-Y). Self-questionnaire assessing anxiety-status (AE) reflecting the current emotional state and anxiety-trait (AT) reflecting the usual emotional state. Total score 20-80.
Change in depression since baseline between groups | Day 28
  Beck Depression Inventory (BDI). The total score is obtained by adding the scores of the 13 items. This score will be between 0 and 63. The higher the score, the more depressed the subject is.
Change in quality of life since baseline | Day 28
  Dysfunctional Beliefs and Attitudes about Sleep - 16 (DBAS-16). This self-questionnaire is composed of 16 items: Perceived consequences of insomnia (5 items), Worry/impotence about insomnia (6 items), Sleep expectations (2 items), Medication (3 items). The global score is an average of the scores of each item, ranging from 0 to 10. The higher the score, the more dysfunctional beliefs and attitudes about sleep
Use of hypnotic drugs between groups | Day 28
  Yes/no for each type
Use of anxiolytic drugs between groups | Day 28
  Yes/no for each type
Dose of any hypnotic drugs taken between groups | Day 28
Dose of any anxiolytic drugs taken between groups | Day 28
Completion of therapeutic education sessions of patients in the therapeutic education group | Day 28
  Yes/no
Length of workshops in the therapeutic education group | Day 28
  Minutes
Problems encountered during workshops of patients in the therapeutic education group | Day 28
  Descriptive list made by investigator
Patient-reported reason for refusal to participate in the therapeutic education group | Day 28
  Descriptive list of reasons given by the patient
Improvement in chronic insomnia between groups | Month 4
  Change in Insomnia Severity Index (ISI) score (Score between 0 - 28) from inclusion
Change in anxiety since baseline between groups | Month 4
  State-Trait Anxiety Inventory (STAI-Y). Self-questionnaire assessing anxiety-status (AE)
Change in depression since baseline between groups | Month 4
  Beck Depression Inventory (BDI). The total score is obtained by adding the scores of the 13 items. This score will be between 0 and 63. The higher the score, the more depressed the subject is.
Change in quality of life since baseline | Month 4
  Dysfunctional Beliefs and Attitudes about Sleep - 16 (DBAS-16). This self-questionnaire is composed of 16 items: Perceived consequences of insomnia (5 items), Worry/impotence about insomnia (6 items), Sleep expectations (2 items), Medication (3 items). The global score is an average of the scores of each item, ranging from 0 to 10. The higher the score, the more dysfunctional beliefs and attitudes about sleep

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Abril, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de NIMES, Nîmes, France